CLINICAL TRIAL: NCT03992157
Title: Evaluation of Ambulatory ECG Telemetry for the Early Detection of Atrial Fibrillation During Hospital Assessment of Cerebral Infarction
Acronym: TELEMETRIE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Medical practices have evolved and are not conform with the study procedure. Actually, all patients receive an ambulatory ECG telemetry monitoring
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-38
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Cerebral Infarction
Keywords: stroke; ECG; telemetry; atrial fibrillation
MeSH Terms: conditions — Cerebral Infarction; Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- holter-ECG (Experimental): Implementation of an ECG Holter during hospitalisation patient.
  Interventions: Device: ECG telemetry
- Crontrole (No Intervention): No implementation of an ECG Holter

INTERVENTIONS:
Device: ECG telemetry — ECG telemetry (holter ECG) is a portable case - attached to the belt or around the neck - connected to 6 electrodes placed on the skin next to the heart. They are worn by patients during their stay in hospital
  Arms: holter-ECG

SUMMARY:
The aim of the study is to show that an ambulatory ECG telemetry monitoring of some patients hospitalized for cerebral infarction increases the frequency of the diagnosis of atrial fibrillation, cause of their stroke, and reinforces the protection against recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Diagnosis of transient ischemic or cerebral accident
* Absence of etiological orientation after the initial assessment (including at least cerebral MRI, angiography of the supra aortic trunks by CT or MRI, echocardiography with search for patent foramen ovale, standard biology)
* Affiliated to a social security system.
* Having given no opposition to participation in research

Exclusion Criteria:

* AF known or diagnosed during stay in USINV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic impact of outpatient ECG telemetry | 6 months
  Percentage of patients hospitalized for cerebral infarction and with a diagnosis of atrial fibrillation allowed by the use of ambulatory ECG telemetry.

SECONDARY OUTCOMES:
Identification of prognostic factors to identify de novo atrial fibrillation | 6 months
  Retrospective evaluation of prognostic criteria (clinical data, biomarkers, abdominal MRI) in patients with a diagnosis of AF
Evaluate the therapeutic impact (prescription anticoagulant) at the end of hospitalisation | 6 months
  Percentage of patients on anticoagulation at the end of hospitalisation
Evaluate the benefit on the recurrence rate of cerebral infarction after the exit of the service | 3 months
  Percentage of IC recurrence in the department and within 3 months of the IC diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lapergue, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No